CLINICAL TRIAL: NCT02181075
Title: A Proof of Concept Study to Investigate the Feasibility of Targeted Release of Doxorubicin From Lyso-thermosensitive Liposomal (LTSL) Doxorubicin (ThermoDox®) Using Focused Ultrasound in Patients With Primary or Secondary Liver Tumours
Brief Title: Targeted Chemotherapy Using Focused Ultrasound for Liver Tumours
Acronym: TARDOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Imunon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_040; 2014-000514-61 (EudraCT Number)
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2018-11

CONDITIONS: Liver Tumour
Keywords: ThermoDox; High Intensity Focused Ultrasound; Lyso thermosensitive Liposomal; Non invasive drug delivery; Hepatic metastatic disease; Liver tumour(s); Targeted Release of Chemotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Parts I and II of the study were not randomised, and both Parts of the study are detailed further in the published protocol summary, detailed in References section. After a minimum of 5 patients were treated in Part 1 (Arm 1), Part 2 (Arm 2) of the study could be opened.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part I (Experimental): All participants in Part I received:
  Pre-LTLD Biopsy of Target Liver Tumour ThermoDox® (LTLD) Post-LTLD Biopsy of Target Liver Tumour Focused Ultrasound of Target Liver Tumour Thermometry of Target Tumour Post-LTLD+FUS (Post-FUS) Biopsy of Target Liver Tumour
  Part I of the study was designed to identify optimal focused ultrasound (FUS) exposure parameters for a range of tumour locations within the liver, using real-time thermometry data from an implanted thermometry device (a thermistor or thermocouple). Plasma and biopsy samples of the target liver tumour were taken pre-LTLD, post-LTLD and post-LTLD+FUS.
  Interventions: Drug: ThermoDox® (LTLD); Device: Focused Ultrasound of Target Liver Tumour; Diagnostic Test: Pre-LTLD Biopsy of Target Liver Tumour; Diagnostic Test: Post-LTLD Biopsy of Target Liver Tumour; Diagnostic Test: Post-LTLD+FUS (Post-FUS) Biopsy of Target Liver Tumour; Device: Thermometry of Target Tumour
- Part II (Experimental): All participants in Part II received:
  ThermoDox® (LTLD) Focused Ultrasound of Target Liver Tumour Post-LTLD Biopsy of Target Liver Tumour
  Following a minimum of 5 Part I cases, and subject to Trial Management Group approval, Part II of the study was opened to run in parallel to Part I. Part II did not require implantation of a thermometry device, and instead used predictions from Part I data to set the FUS parameters. Targeted drug delivery in Part II thus proceeded completely non-invasively, and this part of the study was designed to more closely reflect how the therapy might be implemented in routine clinical practice. Plasma samples were taken pre-LTLD, post-LTLD and post-LTLD+FUS. Biopsy samples of the target liver tumour were taken only post-LTLD+FUS.
  Interventions: Drug: ThermoDox® (LTLD); Device: Focused Ultrasound of Target Liver Tumour; Diagnostic Test: Post-LTLD+FUS (Post-FUS) Biopsy of Target Liver Tumour

INTERVENTIONS:
Drug: ThermoDox® (LTLD) — ThermoDox® (LTLD) infusion at a dose of 50mg/m2 whilst under general anaesthetic during intervention (Day 1)
  Other Names: Lyso-thermosensitive Liposomal Doxorubicin
Device: Focused Ultrasound of Target Liver Tumour — Whilst the ThermoDox® was circulating in the blood stream, the JC200 Therapeutic Ultrasound device was used to induce mild hyperthermia in a single (region of) a target liver tumour.
Diagnostic Test: Pre-LTLD Biopsy of Target Liver Tumour
  Arms: Part I
Diagnostic Test: Post-LTLD Biopsy of Target Liver Tumour
  Arms: Part I
Diagnostic Test: Post-LTLD+FUS (Post-FUS) Biopsy of Target Liver Tumour
Device: Thermometry of Target Tumour — A clinically approved thermistor or thermocouple was placed in the target liver tumour for real-time thermometry.
  Arms: Part I

SUMMARY:
This proof of concept study proposes targeted delivery of a broad-spectrum cytotoxic agent (doxorubicin), via a specially formulated LTSL (ThermoDox®) activated by mild hyperthermia, by using focused ultrasound (FUS), to achieve enhanced intra-tumoural doxorubicin concentrations for the same systemic dose.

Adult patients with incurable confirmed hepatic primary or secondary tumours received a single cycle of LTLD, followed by ultrasound-mediated hyperthermia to a single target liver tumour. The primary endpoint relates to evidencing enhanced delivery of doxorubicin from LTLD at the target tumour site, by comparing intratumoural concentrations of the drug before and after focused ultrasound (FUS) exposure.

DETAILED DESCRIPTION:
To date, purely pharmacological approaches have failed to address what is essentially a threefold challenge: (i) to deliver therapeutically significant concentrations of active agents to the tumour vasculature while minimizing off target effects; (ii) to release the therapeutic agent 'on-demand' at the target site; and, (iii) to improve the distribution and spread of the therapeutic agent against the intra-tumoural pressure gradient in order to achieve a therapeutically relevant concentration throughout the tumour.

Recent pre-clinical studies performed at Oxford using ThermoDox® released using FUS has shown that increased uptake at the target site is achievable. Hence there is great promise in using this combination therapy to achieve increased tumour uptake and local dose for the equivalent dose of doxorubicin used in systemic chemotherapy for human subjects, which has a well established and safe toxicity profile. The first extracorporeal FUS device in Europe was used for a study performed at Oxford between 2002 and 2004.

This single centre trial was sponsored by the University of Oxford. The recruiting study site was Oxford University Hospitals NHS Trust, where there is extensive clinical FUS experience.

The study is split into two parts. Part I identified optimal FUS exposure parameters for a range of patient BMIs and tumour locations within the liver using real time thermometry data from an implanted thermistor. After at least 5 and no more than 14 participants have had the intervention using real-time thermometry, data was reviewed by the Trial Management Group (TMG) to confirm readiness to proceed without real-time thermometry. Part II, which did not require thermistor implantation, is designed to reflect how the therapy would be implemented in clinical practice.

Participants received treatment for 1 day and are followed up for 30 days. All evaluable participants from both Part I and Part II were included in the endpoint analysis. Doxorubicin concentrations were directly determined from tissue biopsies of the target tumour, using a Good Laboratory Practice-validated high performance liquid chromatography (HPLC) assay, based on previously published methods.

If this study demonstrates successful targeted drug delivery in human subjects using LTSLs released by mild-hyperthermia, this could potentially transform the future of chemotherapy in clinical practice; targeted therapy using LTSLs containing other chemotherapeutic agents triggered non-invasively by mild hyperthermia could be applied to any solid organ cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed advanced solid tumour with liver metastasis suitable for intervention (as assessed by ultrasound or other radiological methods). In addition confirmed primary liver tumours (hepatocellular carcinoma or cholangiocarcinoma) can be included.
* Will have progressed or remained stable on conventional chemotherapy.
* Male or Female, Age ≥ 18 years.
* Have life expectancy of ≥ 3 months.
* Left Ventricular Ejection Fraction (LVEF) ≥ 50% on echocardiogram.
* Have not received radiotherapy to the target area within the preceding 12 months.
* A World Health Organisation (WHO) performance status of ≤ 1 - Able and willing to give written informed consent, indicating that they are aware of the investigational nature of this study and potential risks, and able to comply with the protocol for the duration of the study, including scheduled follow-up visits and examinations.

Exclusion Criteria:

* Have surgery or other procedure requiring general anaesthesia planned to be undertaken during the period of the study.
* Have serious illnesses including, but not limited to, congestive heart failure (NYHA class III or IV functional classification); life threatening cardiac arrhythmia; or myocardial infarction or cerebral vascular accident within the last 6 months.
* Have on going significant infection (chest, urine, blood, intra-abdominal).
* Have uncontrolled diabetes.
* Have Have received a life-time dose of doxorubicin > 450 mg/m2 or a life-time dose of epirubicin > 900 mg/m2 or any dose of both.
* Pregnant or breast-feeding. In women of childbearing potential, a negative pregnancy test (serum) is required within 30 days prior to study intervention.
* Female participants of child bearing potential and male participants whose partner is of child bearing potential who are not willing to practice an acceptable form of contraception (i.e. oral contraceptive, diaphragm, cervical cap, condom, surgical sterility) during the study and for 6 months thereafter. Women whose partner has or men who have undergone a vasectomy must use a second form of birth control.
* Have any known allergic reactions to any of the drugs or liposomal components or intravenous imaging agents to be used in this study.
* Have portal or hepatic vein tumour invasion/thrombosis.
* Inadequate haematological and biochemical function (as listed in protocol)
* Have contraindications to receiving doxorubicin including prior sensitivity (rash, dyspnoea, wheezing, urticarial or other symptoms) attributed to anthracyclines or other liposomal drugs.
* Use of chemotherapy or of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the intervention.
* Have medically significant active infection.
* Have Child-Pugh Class C liver disease, or Class A-B with encephalopathy and/or refractory ascites.
* Documented HIV positive.
* Documented diagnosis of haemochromatosis.
* Documented history of contrast-induced nephropathy.
* Have any of the following contraindications for liver biopsy:

  1. Suspected liver haemangioma or other vascular tumour
  2. Tense ascites
  3. Known cystic liver disease*
  4. Extra-hepatic biliary obstruction*

     (* Relative contraindications only and may be non-exclusive at discretion of the study team)
* Other medical or psychiatric conditions or laboratory abnormalities that the investigator considers would make the patient a poor trial candidate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Middleton, PhD, FRCP, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Key patient data with tumour characteristics is available in the Lancet Oncology clinical paper (https://doi.org/10.1016/S1470-2045(18)30332-2).

REFERENCES:
- [Background] Lyon PC, Griffiths LF, Lee J, Chung D, Carlisle R, Wu F, Middleton MR, Gleeson FV, Coussios CC. Clinical trial protocol for TARDOX: a phase I study to investigate the feasibility of targeted release of lyso-thermosensitive liposomal doxorubicin (ThermoDox(R)) using focused ultrasound in patients with liver tumours. J Ther Ultrasound. 2017 Nov 2;5:28. doi: 10.1186/s40349-017-0104-0. eCollection 2017. PMID 29118984
- [Background] Kreb DL, Bosscha K, Ernst MF, Rutten MJ, Jager GJ, van Diest PJ, van der Linden JC. Use of cytokeratin 8 immunohistochemistry for assessing cell death after radiofrequency ablation of breast cancers. Biotech Histochem. 2011 Dec;86(6):404-12. doi: 10.3109/10520295.2010.517473. Epub 2010 Oct 18. PMID 20950219
- [Result] Lyon PC, Gray MD, Mannaris C, Folkes LK, Stratford M, Campo L, Chung DYF, Scott S, Anderson M, Goldin R, Carlisle R, Wu F, Middleton MR, Gleeson FV, Coussios CC. Safety and feasibility of ultrasound-triggered targeted drug delivery of doxorubicin from thermosensitive liposomes in liver tumours (TARDOX): a single-centre, open-label, phase 1 trial. Lancet Oncol. 2018 Aug;19(8):1027-1039. doi: 10.1016/S1470-2045(18)30332-2. Epub 2018 Jul 11. PMID 30001990
- [Result] Gray MD, Lyon PC, Mannaris C, Folkes LK, Stratford M, Campo L, Chung DYF, Scott S, Anderson M, Goldin R, Carlisle R, Wu F, Middleton MR, Gleeson FV, Coussios CC. Focused Ultrasound Hyperthermia for Targeted Drug Release from Thermosensitive Liposomes: Results from a Phase I Trial. Radiology. 2019 Apr;291(1):232-238. doi: 10.1148/radiol.2018181445. Epub 2019 Jan 15. PMID 30644817
- See also: Cancer Research UK Summary of TARDOX Trial & Results — https://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-study-looking-at-targeting-chemotherapy-to-the-liver-using-focused-ultrasound-tardox

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 patients were recruited (6 to Part I of the study and 4 to Part II of the study).
  Patients required at least one liver tumour accessible to ultrasound. Full screening criteria are available from ClinicalTrials.gov or the published protocol summary, both detailed in the References section.
Groups:
- Part I (Patients Enrolled Between March 2015-April 2017): Part I of the study was designed to identify optimal focused ultrasound (FUS) exposure parameters for a range of tumour locations within the liver, using real-time thermometry data from an implanted thermometry device (a thermistor or thermocouple). Patients in Part I receive a single cycle of Lyso- Thermosensitive Liposomal Doxorubicin (LTLD, ThermoDox®) intravenously, at a dose of of 50 mg/m2. After a minimum of five patients have received the Part I intervention with real-time thermometry, data was reviewed by the Trial Management Group (TMG) to confirm readiness to proceed without real-time thermometry in Part II of the study. Plasma and biopsy samples of the target liver tumour were taken pre-LTLD, post-LTLD and post- LTLD+FUS.
  Parts I and II of the study were not randomised, and both Parts of the study are detailed further in the published protocol summary (https://doi.org/10.1186/s40349-017-0104-0).
- Part II (Patients Enrolled Between June 2016-Feb 2017): Following a minimum of 5 Part I cases, and subject to Trial Management Group approval, Part II of the study was opened to run in parallel to Part I. Part II did not require implantation of a thermometry device, and instead used predictions from Part I data to set the FUS parameters. Targeted drug delivery in Part II thus proceeded completely non-invasively, and this part of the study was designed to more closely reflect how the therapy might be implemented in routine clinical practice.
  Plasma samples were taken pre-LTLD, post-LTLD and post-LTLD+FUS. Biopsy samples of the target liver tumour were taken only post-LTLD+FUS.
  Parts I and II of the study are not randomised, and both Parts of the study are detailed further in the published protocol summary (https://doi.org/10.1186/s40349-017-0104-0).
Period: Overall Study
Arm/Group | Part I (Patients Enrolled Between March 2015-April 2017) | Part II (Patients Enrolled Between June 2016-Feb 2017)
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part I: Arm I Patients
- Part II: Arm II Patients
- Total: Total of all reporting groups
Arm/Group | Part I | Part II | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 4 | 10
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.73 (1.60) | 29.13 (5.52) | 26.49 (4.09)

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Total Intratumoral Doxorubicin in Liver Tumour (Biopsies) Following Targeted Release of Doxorubicin From ThermoDox® ('Drug') Using Mild Hyperthermia Generated Non-invasively by Focused Ultrasound (FUS)
Description: Analytical chemistry (High Performance Liquid Chromatography) for total doxorubicin (including both released and unreleased forms) was performed on section of intratumoral biopsy samples in Good Clinical Practice Laboratory, using a validated assay.
  Doxorubicin concentration was evaluated in biopsy samples both post-LTLD and post-LTLD+FUS.
  Tumour samples were not analysed same day and were frozen at -80^oC for subsequent analysis. Required to evaluate the primary endpoint.
Time Frame: Post-intervention sample (Day 1) compared to pre-intervention sample (Day 1)
Measure: Mean (Standard Deviation); unit: ug/g of total doxorubicin(tumour biopsy)
Groups:
- Part I (Patients Enrolled Between March 2015-April 2017): Part I of the study was designed to identify optimal focused ultrasound (FUS) exposure parameters for a range of tumour locations within the liver, using real-time thermometry data from an implanted thermometry device (a thermistor or thermocouple). Patients in Part I receive a single cycle of Lyso-Thermosensitive Liposomal Doxorubicin (LTLD, ThermoDox®) intravenously, at a dose of of 50 mg/m2. After a minimum of five patients have received the Part I intervention with real-time thermometry, data was reviewed by the Trial Management Group (TMG) to confirm readiness to proceed without real-time thermometry in Part II of the study. Plasma and biopsy samples of the target liver tumour were taken pre-LTLD, post-LTLD and post-LTLD+FUS.
  Parts I and II of the study were not randomised, and both Parts of the study are detailed further in the published protocol summary (https://doi.org/10.1186/s40349-017-0104-0).
Arm/Group | Part I (Patients Enrolled Between March 2015-April 2017) | Part II (Patients Enrolled Between June 2016-Feb 2017)
Number analyzed (Participants) | 6 | 4
ug/g of total doxorubicin(tumour biopsy)
  Pre-FUS Intratumoural Doxorubicin Concentration | 2.34 (0.93) | 2.34 (0.93)
  Post-FUS Intratumoural Doxorubicin Concentration | 7.74 (4.09) | 9.8 (8.12)
Statistical Analysis 1: Comparison: Part I (Patients Enrolled Between March 2015-April 2017); A paired t-test was used for Part I (Arm 1) only. Analysis only applies to Part I (Arm 1) because only this study arm has matched Post-LTLD (i.e. post-drug alone) and Post-LTLD+FUS biopsy samples obtained from the same liver tumours before and after targeted drug delivery. In Part II of the study design in which drug delivery occurred completely non-invasively, no Post-LTLD tissue sample is obtained and only a single tumour biopsy is obtained following drug delivery (Post-LTLD+FUS); Test type: Superiority; p = 0.024, t-test, 2 sided — Not adjusted for multiple comparisons. A priori threshold < 0.05; 95% confidence interval (CI)

2. Primary Outcome: Patients Demonstrating >Two-fold Increase in the Amount of Intratumoural Doxorubicin Before and After Focused Ultrasound
Description: To satisfy the primary endpoint, a demonstrable two-fold increase in*, or value exceeding 10μg/g of, the concentration of intra-tumoural doxorubicin at the treated tumour site following FUS-induced mild hyperthermia, was required in at least 50% of evaluable participants.
  * As per the a priori protocol design, in Part II the biopsy prior to FUS-induced mild hyperthermia is not performed and therefore the average value for all evaluable tumours receiving intervention in Part I is used as a comparison for the two-fold increase from pre-FUS to post-FUS biopsy.
Time Frame: Post-LTLD+FUS sample (Day 1) compared to Post-LTLD sample (Day 1)
Measure: Count of Participants; unit: Participants
Groups:
- Part I (Patients Enrolled Between March 2015-April 2017): Arm 1 - see above
- Part II (Patients Enrolled Between June 2016-Feb 2017): Arm 2 - see above
Arm/Group | Part I (Patients Enrolled Between March 2015-April 2017) | Part II (Patients Enrolled Between June 2016-Feb 2017)
Number analyzed (Participants) | 6 | 4
Participants | 4 | 3

3. Secondary Outcome: (Part I Only) Achievement of Satisfactory Hyperthermia Within the Target Liver Tumour for a Range of Participant Body Mass Indices (BMIs) and Tumour Locations Within the Liver (Optimal FUS Exposure Parameters)
Description: Achievement of hyperthermia in the target liver tumour, as determined by real-time thermometry obtained by an indwelling thermometry device.
  For success, sustained and controlled hyperthermia is required in the target tumour, consequent with drug release (in excess of 39.5^oC). Real time thermometry plots for each Part I patient are available in the key Lancet Oncology publication, details available in the References section.
Time Frame: Real-time thermometry monitoring during intervention (Day 1)
Population: In Part II there was no real-time thermometry and this endpoint only applies to Part I patients.
Measure: Count of Participants; unit: Participants
Groups:
- Part I (July 2014-July 2017): Part I of the study was designed to identify optimal focused ultrasound (FUS) exposure parameters for a range of tumour locations within the liver, using real-time thermometry data from an implanted thermometry device (a thermistor or thermocouple). Patients in Part I receive a single cycle of Lyso-Thermosensitive Liposomal Doxorubicin (LTLD, ThermoDox®) intravenously, at a dose of of 50 mg/m2. After a minimum of five patients have received the Part I intervention with real-time thermometry, data was reviewed by the Trial Management Group (TMG) to confirm readiness to proceed without real-time thermometry in Part II of the study. Plasma and biopsy samples of the target liver tumour were taken pre-LTLD, post-LTLD and post-LTLD+FUS.
  Parts I and II of the study were not randomised, and both Parts of the study are detailed further in the published protocol summary (https://doi.org/10.1186/s40349-017-0104-0).
- Part II (May 2016-July 2017): Following a minimum of 5 Part I cases, and subject to Trial Management Group approval, Part II of the study was opened to run in parallel to Part I. Part II did not require implantation of a thermometry device, and instead used predictions from Part I data to set the FUS parameters. Targeted drug delivery in Part II thus proceeded completely non-invasively, and this part of the study was designed to more closely reflect how the therapy might be implemented in routine clinical practice.
  Plasma samples were taken pre-LTLD, post-LTLD and post-LTLD+FUS. Biopsy samples of the target liver tumour were taken only post-LTLD+FUS. Parts I and II of the study are not randomised, and both Parts of the study are detailed further in the published protocol summary (https://doi.org/10.1186/s40349-017-0104-0).
Arm/Group | Part I (July 2014-July 2017) | Part II (May 2016-July 2017)
Number analyzed (Participants) | 6 | 0
Participants | 5 |

4. Secondary Outcome: Persistence of Cell Viability Stain Post-LTLD+FUS
Description: Post-LTLD+FUS tissue from the targeted liver tumours was obtained by biopsy at the time of the intervention, between 24/03/2015 and 29/03/2017. Cytokeratin-8 (CK-8) is a cell viability marker which if present, demonstrates lack of ablative cell death by any ablative modality, including FUS.
  Not all histological cell types express CK8, thus if the Post-LTLD+FUS it may either indicate:
  i) Non-CK8 expression ii) Thermal ablation and consequent cell death.
  Note there was uncertainty about CK8 expression of individual patient tumours prior to recruitment. In this study if the Post-LTLD+FUS tissue shows specific cellular CK8 cellular staining, then it demonstrates that i) the tumour is CK8+, and, ii) the tumour was not instantaneously thermally ablated and any subsequent cell death is likely due to drug delivery/chemo-ablation.
  For more information see key TARDOX Lancet Oncology publication and Cytokeratin 8 reference (both detailed in References section).
Time Frame: Tissue obtained on day of intervention (Day 1). All CK8 cell viability staining was performed within 2 months of sampling.
Population: 5/6 Part I patients and 4/4 Part II patients had tissue which was analysable for CK-8. The Outcome Measure Data Table demonstrates the number of patients from each arm having CK-8 positive tumour biopsy samples post-LTLD+FUS, indicating lack of thermal ablation (which is consistent with desired hyperthermia rather than undesirable FUS ablation).
Measure: Count of Participants; unit: Participants
Arm/Group | Part I (Patients Enrolled Between March 2015-April 2017) | Part II (Patients Enrolled Between June 2016-Feb 2017)
Number analyzed (Participants) | 5 | 4
Participants | 5 | 3

5. Secondary Outcome: Patients With Significant (Grade 3-5) Adverse Event(s) Deemed Related to ThermoDox (LTLD)
Description: Adverse Events are listed separately in the subsequent results, but were also specified as a secondary endpoint in the a priori protocol and thus significant events are summarised here.
  'Definitely' or 'Probably' related events are included.
Time Frame: Up to 30 days post-intervention (Day 1-30)
Measure: Count of Participants; unit: Participants
Arm/Group | Part I (Patients Enrolled Between March 2015-April 2017) | Part II (Patients Enrolled Between June 2016-Feb 2017)
Number analyzed (Participants) | 6 | 4
Participants | 3 | 4

6. Secondary Outcome: Patients With Significant (Grade 3-5) Adverse Event(s) Deemed Related to FUS Procedure
Description: as for outcome 5
Time Frame: Up to 30 days post-intervention (Day 1-30)
Measure: Count of Participants; unit: Participants
Arm/Group | Part I (Patients Enrolled Between March 2015-April 2017) | Part II (Patients Enrolled Between June 2016-Feb 2017)
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Safety and toxicity reported according to NCI CTCAE v4. Adverse events were recorded at day 1 and at approximately 2 and 4 weeks post-intervention following a clinical review.
Arm/Group | Part I (Patients Enrolled Between March 2015-April 2017) | Part II (Patients Enrolled Between June 2016-Feb 2017)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/4
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I (Patients Enrolled Between March 2015-April 2017) (N=6) | Part II (Patients Enrolled Between June 2016-Feb 2017) (N=4)
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Confusion (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I (Patients Enrolled Between March 2015-April 2017) (N=6) | Part II (Patients Enrolled Between June 2016-Feb 2017) (N=4)
Dysphonia (Surgical and medical procedures) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Fatigue or Lethargy (General disorders) | 4 | 2
Nausea (General disorders) | 2 | 2
Abdominal Pain (General disorders) | 1 | 2
Decreased appetite (General disorders) | 2 | 1
Malaise (General disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Constipation (General disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain or discomfort (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Key Lancet Oncology paper (detailed in References section) addresses these limitations:

1. Laboratory limitations not detailed e.g. under/over estimates
2. Tertiary endpoints not presented

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT02181075/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT02181075/SAP_001.pdf